CLINICAL TRIAL: NCT01385241
Title: Feasibility of a Stigma Reduction Intervention for HIV-infected Women
Brief Title: Feasibility of a Stigma Reduction Intervention for Human Immunodeficiency Virus (HIV)-Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00028044; 1R21NR012415-01A1 (NIH)
Record Dates: First submitted 2011-06-14; First posted 2011-06-30 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Human Immunodeficiency Virus (HIV); Self-efficacy; Self-esteem
Keywords: Human Immunodeficiency Virus (HIV); Stigma; Safe disclosure of seropositive status; HIV positive women; Self-efficacy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Received video intervention (Experimental): The group of women who received an Ipod Touch with the video loaded onto it and told to view it at least once a week for the first 4 weeks, and as often as desired in weeks 5-12.
  Interventions: Behavioral: Ipod video
- Did not receive video (No Intervention): This group does not receive the video intervention during the study period, and will complete surveys at baseline, 30 days and 90 days for comparison to the intervention group.

INTERVENTIONS:
Behavioral: Ipod video — This group will be asked to watch the video on their Ipod Touch in its entirety at least once per week during the first four weeks of the study, and as often as desired in weeks 5-12. The participants will be asked to record the times viewed and their feelings/comments in a viewing log, and will be given surveys at 30 and 90 days.
  Arms: Received video intervention

SUMMARY:
The purpose of this study is to test the feasibility of a stigma reduction intervention in Human Immunodeficiency Virus(HIV)-positive women using a video of first-person narratives delivered via personal Ipod Touch.

DETAILED DESCRIPTION:
Nearly 30 years into the Acquired Immune Deficiency Syndrome (AIDS) epidemic, stigma is still hampering efforts to stop its spread. Human Immunodeficiency Virus(HIV)-infected women are particularly vulnerable to both perceived and enacted stigma, which together are referred to as internalized stigma. As the demographic face of HIV infection in the US has changed from being largely a disease of gay white men to one of poor minority women, the debilitating effects of stigma have worsened. It has a profound impact on prevention and treatment efforts; women with HIV infection may be fearful of insisting that their sexual partners wear condoms because of the possibility that this may signal their serostatus, and they may not want to take antiretroviral medications in front of others, fearing that people may ask questions about their pills and the reasons for taking them. The effects of stigma include a cascade of other negative outcomes as well, including poor self-esteem and self-efficacy, especially self-efficacy for disclosure and for coping. Yet it is nearly impossible to intervene with those who stigmatize others because this group is often as broad as the general public, and they may not be interested in an intervention. Therefore, the best approach may be to work with women who are experiencing stigma, in an effort to decrease stigma, improve self-esteem and coping self-efficacy, and facilitate safe disclosure. To date, there have been few interventions to help HIV-infected women deal with stigma. One option would be a video converted to an Moving Picture 4 (MP4) file that can be viewed on an iPod Touch, a small portable viewing device, allowing the woman privacy and safety in viewing. Barroso (primary investigator on the proposed study) assisted in the creation of a video on stigma for women with HIV infection, based on the results of a qualitative metasynthesis. The 45-minute video presents vignettes about five seropositive women and the ways in which stigma has impacted their lives. The primary aim of the proposed study is to assess the feasibility, acceptability and utility of implementing this low-cost, technologically delivered intervention to mitigate the negative effects of HIV-related stigma on seropositive women. The secondary aim is to compare outcomes across time in women who receive the stigma intervention with those of a control group receiving usual care at baseline, 30, and 90 days, and to determine effect sizes for a larger definitive study to test the efficacy of this intervention in reducing internalized stigma, improving coping self-efficacy and self-esteem, and facilitating safe disclosure in HIV-infected women. The investigators believe that this intervention is innovative because they are the first investigators to propose using a video, developed from the findings of a metasynthesis of studies about stigma as it is experienced by HIV-infected women, for this purpose. It is also innovative in the use of a portable viewing device which will allow the women to safely and privately view the video. The investigators further believe that this intervention has the potential to make a significant impact, at a low cost in terms of money and personnel time, in mitigating stigma.

ELIGIBILITY:
Inclusion Criteria:

* speaks, understands, and reads English
* Scores over 40 on Internalized Human Immunodeficiency Virus (HIV) Stigma Scale
* HIV positive
* mentally competent to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing a stigma reduction intervention among Human Immunodeficiency Virus (HIV)-infected women | 90 days
  We will test whether the use of an Ipod Touch video intervention is feasible in this study population by comparing baseline data with data collected at 30 days into the intervention and upon completion of the intervention at 90 days.

SECONDARY OUTCOMES:
Acceptability of the use of a portable device to deliver a video intervention among Human Immunodeficiency Virus(HIV)-infected women | 90 days
  We will test whether the means and the method employed to deliver this intervention are acceptable to the study population through the collection of qualitative data at 30 days and 90 days.
Utility of the use of a portable media device to deliver stigma-reduction intervention among Human Immunodeficiency Virus(HIV)-infected women | 90 days
  We will test whether the intervention method is useful to the study population in achieving the desired outcome by measuring feelings of stigma at baseline, 30 days and 90 days and assessing positive change.
Change from baseline in levels of internalized stigma | 90 days
  We will test whether this intervention reduces the level of internalized stigma experienced by Human Immunodeficiency Virus(HIV)-positive women, comparing baseline levels with levels at 30 days and 90 days.
Change from baseline in levels of coping self-efficacy | 30 days, 90 days
  We will test whether this study increases the coping skills and belief in ability to cope in the women who receive it.
Change in safe disclosure behaviors from baseline | 90 days
  Though they were not expressly told to disclose their status as a part of this study, we would like to find out whether this video inspires women to disclose their status to family members, sexual partners, and other support people whom they deem to be safe and trustworthy confidantes.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Barroso, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University clinics, Henderson, North Carolina, United States